CLINICAL TRIAL: NCT02764099
Title: Testing a Multilevel Preventive Intervention in Youth Courts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Williams, Senior Vice President, National Health Promotion Associates, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R34DA034888 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2016-05-06 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Life Skills Training (Experimental): All youth who consent to participate in the proposed study will 1) complete the youth peer court sanction delivered by the jury of peers (e.g., apologies or essays, restitution, curfew and travel restrictions, counseling, etc.), which will constitute "treatment as usual"; and 2) complete pre, post, and six-month follow-up surveys. Those randomized to the intervention condition (n=280) will participate in the LST program concurrently during the weeks when they serve as peer court jurors.
  Interventions: Behavioral: Life Skills Training

INTERVENTIONS:
Behavioral: Life Skills Training — The Life Skills Training (LST) program is a comprehensive competence enhancement prevention approach that teaches resistance skills while also emphasizing generic personal and social skills training. The LST program content and skills training is delivered to youth participants by trained providers through instruction, demonstration, behavioral rehearsal with feedback and social reinforcement, extended practice through homework assignments, and didactic teaching methods.
  Other Names: LST

SUMMARY:
The proposed research is designed to adapt and test an evidence-based drug abuse prevention approach for use in youth courts among first-time, non-violent, adolescent offenders. The ultimate goal is to reduce the adverse health, legal, and social consequences of youth drug abuse, violence, and delinquency. Planned project activities include conducting: 1) key informant interviews of youth court directors regarding logistical and intervention features of effective youth court programming; and, 2) a randomized controlled efficacy trial of an adapted version of Life Skills Training, an evidence-based drug and violence prevention program. It is anticipated that the findings will provide critical information on implementing evidence-based prevention programs for new populations and settings and will support preparations for a large-scale effectiveness trial in youth peer courts.

DETAILED DESCRIPTION:
Adolescents in under-served, urban communities are disproportionately involved in the juvenile justice system. This early engagement has been shown to be a strong predictor of more serious offenses in adulthood, such that youth involvement in the court system is a significant public health concern. Juvenile justice approaches have traditionally emphasized individualized treatment efforts combined with discipline and punishment. More recently, however, juvenile justice professionals have questioned the adequacy of this approach and are increasingly adopting an asset-based perspective referred to as "positive youth justice" (PYJ). The PYJ approach encourages youth court participants to build upon their existing strengths, while learning and mastering new life skills, through development of pro-social relationships within their peer group, family, and community. These "core assets" are posited to promote the successful entry into young adulthood. For this project, the investigative team will adapt and test a multilevel, multi-component, intervention that has strong potential to reduce substance use and delinquency while correspondingly promoting positive youth justice among youth court participants and staff. The first component of the current project involves interviewing program directors from a representative sample of youth courts throughout the U.S to gain formative feedback about logistical and programming concerns. The second component of the project is designed to promote individual-level change among youth participants and consists of an adapted version of the Life Skills Training (LST) program, an evidence-based drug and violence prevention program which teaches personal self-management skills, social skills, drug refusal skills, and other life skills needed to successfully navigate developmental tasks, increase resilience, and facilitate healthy psycho-social development. Several youth courts have used the Life Skills Training program, suggesting that it meets a perceived need and is feasible in this setting. However, LST has never been rigorously tested in the youth court setting. The proposed research will involve a randomized efficacy trial with 560 adolescents in youth court. The investigative team will examine intervention effects on substance use, delinquent behavior, school performance, and recidivism rates using mixed qualitative (assessment of dosage, fidelity, and provider and participant feedback to determine their impact on program efficacy) and quantitative (survey assessments at pretest, post-test, and six-month follow-up) methods to estimate the effect size of the adapted and combined program. By intervening with both youth court participants and youth court staff, the proposed multilevel intervention can have a broad impact on risk and protective factors at multiple levels of influence. The ultimate goal of this research is to promote the use of an evidence-based prevention approach adapted specifically for implementation in youth courts in order to reduce the adverse consequences of drug abuse, violence, and delinquency among youth offenders.

The specific aims of this project will be to:

1. Conduct key informant interviews with a diverse sample of youth court program coordinators;
2. Conduct expert review of the LST intervention materials to ensure accuracy and appropriateness for the youth court setting and revise appropriately for an efficacy trial;
3. Evaluate the efficacy of the combined youth court intervention (staff training plus LST) in preventing substance use, delinquency and violence, improving hypothesized mediators of intervention effects, including knowledge, attitudes and life skills, and promoting effective youth placements in community settings;
4. Examine the degree to which process variables such as dosage and fidelity moderate intervention effects;
5. Examine all recruitment, incentive, consent, tracking and assessment procedures in preparation for a subsequent national effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for youth participants will include regular participation in youth court activities and informed consent

Exclusion Criteria:

* Exclusion criteria for youth participants will include significant cognitive impairment or severe learning disabilities, as screened by staff at the youth court
* Any previous experience with the intervention program will also exclude adolescents from participating

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 423 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Substance Use Behavior, Intentions, Attitudes and Perceived Norms at Baseline | Pre-test (prior to participating in the first session of the intervention)
  Substance Use Behavior and Intentions: For 13 substance-related items (e.g., alcohol, tobacco, cocaine, methamphetamines, steroids), participants will be asked to indicate frequency of use. Drug Attitudes: Sixteen items will be used to assess participants' attitudes about drug use, perceived characteristics of drug users and the perceived social benefits of drug use. Drug Norms & Knowledge: Normative expectations related to drug use will be assessed including perceived prevalence of drug use among peers and among adults. Friends' and adult substance use will be measured. Drug Refusal Skills will be assessed using five items that measure the ability to resist peer pressure to engage in substance use.
Change in Baseline Substance Use Behavior, Intentions, Attitudes and Perceived Norms at Post-Intervention | Post-test (within 2 weeks of completing final session of the intervention)
  Substance Use Behavior and Intentions: For 13 substance-related items (e.g., alcohol, tobacco, cocaine, methamphetamines, steroids), participants will be asked to indicate frequency of use. Drug Attitudes: Sixteen items will be used to assess participants' attitudes about drug use, perceived characteristics of drug users and the perceived social benefits of drug use. Drug Norms & Knowledge: Normative expectations related to drug use will be assessed including perceived prevalence of drug use among peers and among adults. Friends' and adult substance use will be measured. Drug Refusal Skills will be assessed using five items that measure the ability to resist peer pressure to engage in substance use.
Change in Baseline Substance Use Behavior, Intentions, Attitudes and Perceived Norms at 6-months | 6-month followup (within 6-7 months of completing final session of intervention)
  Substance Use Behavior and Intentions: For 13 substance-related items (e.g., alcohol, tobacco, cocaine, methamphetamines, steroids), participants will be asked to indicate frequency of use. Drug Attitudes: Sixteen items will be used to assess participants' attitudes about drug use, perceived characteristics of drug users and the perceived social benefits of drug use. Drug Norms & Knowledge: Normative expectations related to drug use will be assessed including perceived prevalence of drug use among peers and among adults. Friends' and adult substance use will be measured. Drug Refusal Skills will be assessed using five items that measure the ability to resist peer pressure to engage in substance use.

SECONDARY OUTCOMES:
Aggressive, Violent, and Delinquent Behavior at Baseline | Pre-test (prior to participating in the first session of the intervention)
  Aggressive, violent, and delinquent behaviors will be assessed using the items from the Reactive/Proactive Aggression Scale (RPAS). The RPAS provides respondents with a sequence of aggressive/violent behaviors and prompts them to indicate the frequency of each behavior. Beliefs about aggressive and violent behavior will be measured using the items from the Normative Beliefs about Aggression Scale (NBAS). The 20-item NBAS contains 2 sections: retaliation belief questions and general belief questions, which can be tallied to calculate a measure of total approval of aggression. Delinquent and disciplinary behavioral data will be gathered using the Rochester Youth Development Self-Reported Delinquency Scale, a self-report measure of delinquency and problem behavior developed by the Rochester Youth Development Study.
Change in Baseline Aggressive, Violent, and Delinquent Behavior at Post-Intervention | Post-test (within 2 weeks of completing final session of the intervention)
  Aggressive, violent, and delinquent behaviors will be assessed using the items from the Reactive/Proactive Aggression Scale (RPAS). The RPAS provides respondents with a sequence of aggressive/violent behaviors and prompts them to indicate the frequency of each behavior. Beliefs about aggressive and violent behavior will be measured using the items from the Normative Beliefs about Aggression Scale (NBAS). The 20-item NBAS contains 2 sections: retaliation belief questions and general belief questions, which can be tallied to calculate a measure of total approval of aggression. Delinquent and disciplinary behavioral data will be gathered using the Rochester Youth Development Self-Reported Delinquency Scale, a self-report measure of delinquency and problem behavior developed by the Rochester Youth Development Study.
Change in Baseline Aggressive, Violent, and Delinquent Behavior at 6-months | 6-month followup (within 6-7 months of completing final session of intervention)
  Aggressive, violent, and delinquent behaviors will be assessed using the items from the Reactive/Proactive Aggression Scale (RPAS). The RPAS provides respondents with a sequence of aggressive/violent behaviors and prompts them to indicate the frequency of each behavior. Beliefs about aggressive and violent behavior will be measured using the items from the Normative Beliefs about Aggression Scale (NBAS). The 20-item NBAS contains 2 sections: retaliation belief questions and general belief questions, which can be tallied to calculate a measure of total approval of aggression. Delinquent and disciplinary behavioral data will be gathered using the Rochester Youth Development Self-Reported Delinquency Scale, a self-report measure of delinquency and problem behavior developed by the Rochester Youth Development Study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Williams, Ph.D., Principal Investigator — National Health Promotion Associates

IPD SHARING:
Plan to Share IPD: No